CLINICAL TRIAL: NCT03565770
Title: Assessment of Individual Follow-up by Reference Nurses (Telemedicine Coaching Program) for Type 1 Diabetes Children With Therapy Adjustment Difficulties
Brief Title: Assessment of Individual Follow-up by Coaching Program for Type 1 Diabetes Children
Acronym: DIAB-HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016_65; 2017-A03021-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetes type1
Keywords: child; coaching; telemedicine; nurses; individual follow-up
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care + coaching (Experimental): minor patients with a type 1 diabetes, having therapy adjustment difficulties, receiving individual coaching and usual standard care
  Interventions: Other: individual coaching; Other: Standard care
- Standard care (Sham Comparator): minor patients with a type 1 diabetes, having therapy adjustment difficulties, receiving usual standard care only.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: individual coaching — coaching on the phone or with messages on line twice a month in order to help patients to adjust their insulin doses and fill in their self-assessment test.
  Arms: standard care + coaching
Other: Standard care — completion of the self-assessment test at inclusion, at M6 and M12 for all study participants

SUMMARY:
The purpose of this project is to assess the introduction of an individual follow-up distance coaching (phone and messages on a secure line platform) in order to optimize the health care of type 1 diabetes children with therapy adjustment difficulties. It is a personalized, multi-disciplinary, medical et paramedical. It will consist of an individual coaching for the children and families with therapy adjustment difficulties.

The hypothesis is that the proposed coaching would allow to improve the patient glycemic control not only during this coaching, but also, to bring long lasting improvement following the coaching.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years old when coaching starts.
* Any diabetic patient (girl or boy) who doesn't master the adjustments of the treatment according to the investigator's judgment (non-adaptations of the treatment between 2 consultations or mistakes in adapting the insulin doses, not taking properly into account previous days tendencies, food, or activities) and/or average HbA1c of more than 8% during the last year.
* The patient, his 2 parents or legal representatives all agree to participate in the research
* Absence of justice protection measures
* Good predictable observance of the protocol
* Family can be reached by phone during the coaching timetables working hours or must be listed on the platform line " MyDiabby ".

Exclusion Criteria:

* Non auto-immun diabetes
* Major understanding difficulties from the relatives (difficulties in understanding French or what anticipatory adaptation means)
* The child or parents or legal representatives refuse to participate and to sign a consent
* Contact on the phone or on the platform impossible according to the protocol procedures
* Patient non-registered under Social Security
* Patient under justice protection measures

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Difference between the rate of glycosylated hemoglobin (HbA1c) before randomization (baseline) and the rate of glycosylated hemoglobin after 6 months coaching (measure M6). | at 6 months

SECONDARY OUTCOMES:
Difference between the rate of glycosylated hemoglobin (HbA1c) before randomization (baseline) and the follow-up. | at baseline, at 3 months, at 12 months
Rate of patients presenting at least one bad accident (ketoacidosis and/or severe hypoglycemia) | at 6 months
Patient self-assessment score | at baseline, at 6 months, at 12 months
Capacity of proper adjustment of the treatment: binary variable " yes/no " evaluated to the judgment of the investigator | at baseline, at 6 months, at 12 months
Binary variable attendance = 80% honored appointments | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lefe, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, Lille, France